CLINICAL TRIAL: NCT04643483
Title: A Phase 3, Randomized, Double-Blind, Multicenter Study Including an Active Reference Arm to Evaluate Efficacy, Safety, and Pharmacokinetics of Certolizumab Pegol in Children and Adolescents (6 to 17 Years of Age) With Moderately to Severely Active Crohn's Disease
Brief Title: A Study to Test Efficacy, Safety, and Pharmacokinetics of Certolizumab Pegol in Children and Adolescents With Moderately to Severely Active Crohn's Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD0003
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Crohn's Disease
Keywords: Certolizumab pegol; Cimzia; Phase 3; Crohn's disease; Pediatric; Kids; OHANA; CD
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol; Adalimumab

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 3 parts:
  * Part A will investigate 2 certolizumab pegol (CZP) dosing regimens with the objective of selecting a regimen that provides the highest rate of clinical remission. A cohort of participants will receive adalimumab (ADA) as a reference arm in Part A to assess clinical remission rates at Week 26 in this population. Endoscopic remission at Week 26 will also be evaluated
  * Part B will assess maintenance of clinical remission from Week 26 through Week 52
  * Part C is an optional open-label extension (OLE) of CZP after Part B, and will evaluate the long-term safety of CZP through Week 156
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Certolizumab pegol low dose arm (Experimental): Participants randomized to certolizumab pegol (CZP) who weigh ≥17 kg to <40 kg will receive placebo at Week 0 and a loading dose of 200 mg at Weeks 0, 2, and 4, followed by a maintenance dose of 100 mg CZP subcutaneously (sc) every 2 weeks (Q2W).
  Participants randomized to CZP who weigh ≥40 kg will receive placebo at Week 0 and a loading dose of 400 mg at Weeks 0, 2, and 4, followed by placebo and a maintenance dose of 200 mg CZP sc Q2W.
  Interventions: Drug: Certolizumab pegol; Drug: Placebo
- Certolizumab pegol high dose arm (Experimental): Participants randomized to CZP who weigh ≥17 kg to <40 kg will receive placebo at Week 0 and a loading dose of 200 mg at Weeks 0, 2, and 4, followed by a maintenance dose of 200 mg CZP sc Q2W.
  Participants randomized to CZP who weigh ≥40 kg will receive placebo at Week 0 and a loading dose of 400 mg at Weeks 0, 2, and 4, followed by a maintenance dose of 300 mg CZP sc Q2W.
  Interventions: Drug: Certolizumab pegol; Drug: Placebo
- Adalimumab reference arm (Active Comparator): Participants randomized to adalimumab who weigh ≥17 kg to <40 kg will receive a loading dose of 80 mg at Week 0 and 40 mg at Week 2, followed by a maintenance dose of 20 mg sc Q2W.
  Participants randomized to Adalimumab who weigh ≥40 kg will receive a loading dose of 160 mg at Week 0 and 80 mg at Week 2, 40 mg and placebo at week 4 followed by a maintenance dose of 40 mg sc and placebo Q2W.
  Interventions: Drug: Adalimumab; Drug: Placebo

INTERVENTIONS:
Drug: Certolizumab pegol — * Pharmaceutical form: Solution for injection
  * Route of administration: Subcutaneous
  Subjects will receive certolizumab pegol in a pre-specified sequence during the Treatment Periods.
  Arms: Certolizumab pegol high dose arm; Certolizumab pegol low dose arm
Drug: Adalimumab — * Pharmaceutical form: Solution for injection
  * Route of administration: Subcutaneous
  Subjects will receive adalimumab in a pre-specified sequence during the Treatment Periods.
  Arms: Adalimumab reference arm
Drug: Placebo — * Pharmaceutical form: Solution for injection
  * Route of administration: Subcutaneous
  Subjects will receive placebo in a pre-specified sequence during the Treatment Periods.

SUMMARY:
The purpose of the study is to assess efficacy, safety and tolerability of 2 dose regimens of certolizumab pegol

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 6 to 17 years, inclusive, at the time of signing informed consent/assent
* Participant has been diagnosed with active Crohn's disease (CD) as confirmed by endoscopic examination with/without histological confirmation ≤12 weeks before the Screening Visit
* Participant has moderately to severely active disease despite current treatment
* Participant has an inadequate response or intolerance to conventional therapy
* Participants are certolizumab pegol (CZP) and adalimumab (ADA) naïve

Exclusion Criteria:

* Participant has had an extensive colonic resection, subtotal or total colectomy, diagnosis of short bowel syndrome or a history of >3 small bowel resections
* Participant has had a primary failure (ie, lack of response within the first 12 weeks of treatment) to any anti-Tumor necrosis factor-α agent for treatment of Crohn's disease

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Clinical remission based on total Pediatric Crohn's Disease Activity Index (PCDAI) score ≤10.0 points at Week 26 | Week 26
  Clinical remission is defined as a Pediatric Crohn's Disease Activity Index (PCDAI) score ≤ 10.
  The Pediatric Crohn's Disease Activity Index (PCDAI) consists of 4 domains (laboratory, height/weight, examination, and history) with several assessments that are converted into a total PCDAI score which can range from 0 to 100 points, with a higher score indicating more severe disease activity.

SECONDARY OUTCOMES:
Clinical remission (modified) at Week 26 | Week 26
  Clinical remission (modified) is defined as a Pediatric Crohn's Disease Activity Index (PCDAI) score ≤ 10 and the abdominal pain and stool frequency items in the PCDAI having scores of 0.
  The Pediatric Crohn's Disease Activity Index (PCDAI) consists of 4 domains (laboratory, height/weight, examination, and history) with several assessments that are converted into a PCDAI score which can range from 0 to 100 points, with a higher score indicating more severe disease activity.
Corticosteroid-free clinical remission at Week 26 | Week 26
  Corticosteroid free clinical remission is defined as not taking corticosteroids after tapering, within 4 weeks prior to Week 26, and total PCDAI score ≤10.0 points and the abdominal pain and stool frequency items in the PCDAI having scores of 0 at Week 26.
Clinical response at Week 26 and Week 52 | Week 26; Week 52
  Clinical response is defined as a decrease from Week 0 in Pediatric Crohn's Disease Activity Index (PCDAI) score of ≥ 15 points and a total PCDAI score ≤ 30 points. The Pediatric Crohn's Disease Activity Index (PCDAI) consists of 4 domains (laboratory, height/weight, examination, and history) with several assessments that are converted into a PCDAI score which can range from 0 to 100 points, with a higher score indicating more severe disease activity.
Endoscopic remission at Week 26 | Week 26
  Endoscopic remission is defined as Simple Endoscopic Score for Crohn's Disease [SES-CD] from 0 to 2, with a higher score indicating more disease activity. SES-CD is based on four endoscopic variables (presence and size of ulcers, proportion of surface covered by ulcers, proportion of surface affected by disease, and presence and severity of stenosis). Each of the four SES-CD variables is scored from 0 to 3, with the sum of the scores for each variable ranging from 0 to 15, except for the presence and extent of stenosis, which ranges from 0 to 11, yielding a total SES-CD score of 0-56.
Clinical remission based on total PCDAI score ≤10.0 points at Week 52 | Week 52
  Clinical remission is defined as a Pediatric Crohn's Disease Activity Index (PCDAI) score ≤ 10.
  The Pediatric Crohn's Disease Activity Index (PCDAI) consists of 4 domains (laboratory, height/weight, examination, and history) with several assessments that are converted into a total PCDAI score which can range from 0 to 100 points, with a higher score indicating more severe disease activity.
Clinical remission (modified) at Week 52 | Week 52
  Clinical remission (modified) is defined as a Pediatric Crohn's Disease Activity Index (PCDAI) score ≤ 10 and the abdominal pain and stool frequency items in the PCDAI having scores of 0.
  The Pediatric Crohn's Disease Activity Index (PCDAI) consists of 4 domains (laboratory, height/weight, examination, and history) with several assessments that are converted into a PCDAI score which can range from 0 to 100 points, with a higher score indicating more severe disease activity.
Incidence of serious Treatment Emergent Adverse Event (TEAEs) | From Baseline to the Safety Follow-Up visit (Week 166)
  A Serious Treatment Emergent Adverse Event is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent disability/incapacity
  * Is a congenital anomaly/birth defect
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above
Incidence of TEAEs leading to permanent withdrawal of investigational medicinal product | From Baseline to the Safety Follow-Up visit (Week 166)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org